CLINICAL TRIAL: NCT06000501
Title: An Open-Label Treatment, Investigator-Initiated Study, on the Duration and Efficacy of Azstarys (Serdexmethylphenidate and Dexmethylphenidate) on Adult ADHD Symptoms and Executive Function in Early Evening
Brief Title: Duration and Efficacy of Azstarys on Adult ADHD Symptoms and Executive Function in Early Evening
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Corium, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-01003
Record Dates: First submitted 2023-08-14; First posted 2023-08-21 (Actual); Results first posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Adult Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — serdexmethylphenidate and dexmethylphenidate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Adult ADHD Patients (Experimental): Enrolled participants will begin with a two-week observation stabilization before starting treatment with Azstarys. Participants found to have ≥30% change in their total Adult ADHD Investigator Symptom Rating Scale (AISRS) scores during the two-week observation stabilization period treatment will be discontinued from the study. Remaining participants will be dispensed a three-week supply of Azstarys on a weekly basis.
  Interventions: Drug: Serdexmethylphenidate/dexmethylphenidate

INTERVENTIONS:
Drug: Serdexmethylphenidate/dexmethylphenidate — Azstarys capsules for once-daily oral use for three weeks. Flexible dose starting at 39.2 mg serd-mph/7.8 mg d-mph and moving up to 52.3 mg serd-mph/10.4 mg d-mph.
  Other Names: Azstarys

SUMMARY:
This is a single-site study. One purpose of this trial is to extend the safety and efficacy evidence basis for Azstarys in adults with ADHD. This open-label, treatment study will examine the efficacy of Azstarys on ADHD symptoms using the AISRS 18-item total score on the AISRS-expanded; the Adult ADHD Investigator Symptom Rating Scale. The investigators will also examine Executive Function later in the day (early evening, about 12 hours after first morning dosing).

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-60 years, inclusive at the time of consent
* Able to provide signed informed consent
* Any gender
* Subjects with a current primary DSM-5 diagnosis of ADHD of predominantly inattentive presentation, or combined presentations) as confirmed by the Adult ADHD Clinical Diagnostic Scale (ACDS) Version 1.2.5, Subjects who are not receiving any pharmacological treatment for ADHD must have an AISRS 18 item total score of AISRS expanded of ≥ 28 at screening. Subjects who were previously receiving pharmacological treatment for ADHD at screening must have a minimum total AISRS 18 item of AISRS EXPANDED score of ≥ 22 at screening
* Dysthymia and anxiety disorders in remission but stable on psychiatric medication for three weeks or more at the discretion of principal investigator will be allowed- medication for these disorders to remain constant for the duration of the protocol.
* Subjects who are stimulant naïve.

Exclusion Criteria:

* Known hypersensitivity to serdexmethylphenidate, methylphenidate, or product components.
* Concurrent treatment with a monoamine oxidase inhibitor (MAOI), or use of an MAOI within the preceding 14 days.
* Lifetime bipolar disorder, psychotic disorders, autism, intellectual disability except mood disorders accepted under the inclusion criteria at the discretion of the principal investigator.
* Active suicidality within past year, or history of suicide attempt in past 2 years
* Any history of severe past drug dependence determined by the MINI (i.e., a focus of clinical attention or a cause of substantial social or occupational difficulty)
* Concurrent substance abuse and/or history of substance use within 6 months
* Use of any prescribed benzodiazepine
* Any unstable medical or neurological condition; clinically significant medical abnormalities such as cardiovascular abnormalities, and any chronic condition of the central nervous system.
* Any psychotropic medication usage
* Known nonresponse to MPH treatment
* History of allergic reaction or sensitivity to MPH
* Female of childbearing age, who are breastfeeding, pregnant, planning to be pregnant or men planning to make a woman pregnant during the study or for one-month post study
* PI/clinician discretion

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-07-03 (Actual); Study Completion 2024-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lenard Adler, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
The study protocol, statistical analysis plan, outcome measure results and adverse event data will be made available on ClinicalTrials.gov. IPD will not be shared due to capacity constraints and privacy concerns.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adult ADHD Patients
Started | 29
Completed | 17
Not Completed | 12
Not completed — Screen failure | 3
Not completed — Severe past drug dependence determined by the MINI | 2
Not completed — Physician Decision | 4
Not completed — Positive Urine Drug Test (UDT) | 1
Not completed — Scheduling issues | 2

BASELINE CHARACTERISTICS:
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Change in Expanded Adult ADHD Investigator Symptom Rating Scale (AISRS) Total Score
Description: The expanded AISRS is an 34-item questionnaire assessing symptoms of adult ADHD. Items are ranked on a 4-point Likert scale ranging from 0 (none) to 3 (severe). The total score is the sum of responses and ranges from 0 to 102; higher scores indicate more severe symptoms of ADHD.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 15
score on a scale | 24.1 (7.4)

2. Secondary Outcome: Change in Expanded AISRS - Overall Inattentive (IA) Subscale Score
Description: The expanded AISRS is an 34-item questionnaire assessing symptoms of adult ADHD. The 9-item subscale of the AISRS assessing inattentive symptoms of ADHD. Items are ranked on a 4-point Likert scale ranging from 0 (none) to 3 (severe). The total score is the sum of responses and ranges from 0 to 27; higher scores indicate greater overall inattentive symptoms.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 15
score on a scale | 14.3 (4)

3. Secondary Outcome: Change in Expanded AISRS - Hyperactive/Impulsive (HI) Subscale Score
Description: The expanded AISRS is an 34-item questionnaire assessing symptoms of adult ADHD. The 9-item subscale of the AISRS assessing hyperactive/impulsive symptoms of ADHD. Items are ranked on a 4-point Likert scale ranging from 0 (none) to 3 (severe). The total score is the sum of responses and ranges from 0 to 27; higher scores indicate greater hyperactive/impulsive symptoms.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 15
score on a scale | 9.7 (4.2)

4. Secondary Outcome: Change in Expanded AISRS - Overall Executive Dysfunction (EFD) Subscale Score
Description: The expanded AISRS is an 34-item questionnaire assessing symptoms of adult ADHD. The 9-item subscale of the AISRS assessing executive dysfunction symptoms of ADHD. Items are ranked on a 4-point Likert scale ranging from 0 (none) to 3 (severe). The total score is the sum of responses and ranges from 0 to 27; higher scores indicate greater hyperactive/impulsive symptoms.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 15
score on a scale | 14.5 (5.1)

5. Secondary Outcome: Change in Expanded AISRS - Overall Emotional Control (EC) Subscale Score
Description: The expanded AISRS is an 34-item questionnaire assessing symptoms of adult ADHD. The 9-item subscale of the AISRS assessing emotional control symptoms of ADHD. Items are ranked on a 4-point Likert scale ranging from 0 (none) to 3 (severe). The total score is the sum of responses and ranges from 0 to 27; higher scores indicate greater hyperactive/impulsive symptoms.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 15
score on a scale | 5.3 (4.8)

6. Secondary Outcome: Change in Adult ADHD Self Report Scale (ASRS) Symptom Checklist DSM-5 Expanded Score
Description: The ASRS is a 31-item questionnaire that assesses the frequency of ADHD symptoms over the past 7 days. Items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The ASRS includes several subscales: an Inattentive (IA) subscale (n = 9), a Hyperactive-Impulsive (HI) subscale (n = 9), an Executive Function Deficits (EFD) subscale (n = 9), and an Emotional Dyscontrol (ED) subscale (n = 4). It also yields a total combined ADHD symptom score. The total score is calculated as the sum of all item responses and ranges from 0 to 124, with higher scores indicating greater frequency of ADHD symptoms.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 25.6 (13.7)

7. Secondary Outcome: Change in Adult ADHD Self Report Scale (ASRS) Symptom Checklist Inattentive (IA) Subscale Score
Description: The ASRS is a 31-item questionnaire that assesses the frequency of ADHD symptoms over the past 7 days. Items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The ASRS includes several subscales: an Inattentive (IA) subscale (n = 9), a Hyperactive-Impulsive (HI) subscale (n = 9), an Executive Function Deficits (EFD) subscale (n = 9), and an Emotional Dyscontrol (ED) subscale (n = 4). It also yields a total combined ADHD symptom score. The IA score ranges from 0-36. Higher scores indicating greater symptom severity.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 14.4 (7.6)

8. Secondary Outcome: Change in Adult ADHD Self Report Scale (ASRS) Symptom Checklist Hyperactive (HI) Subscale Score
Description: The ASRS is a 31-item questionnaire that assesses the frequency of ADHD symptoms over the past 7 days. Items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The ASRS includes several subscales: an Inattentive (IA) subscale (n = 9), a Hyperactive-Impulsive (HI) subscale (n = 9), an Executive Function Deficits (EFD) subscale (n = 9), and an Emotional Dyscontrol (ED) subscale (n = 4). It also yields a total combined ADHD symptom score. The HI score ranges from 0-36. Higher scores indicating greater symptom severity.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 11.1 (7.2)

9. Secondary Outcome: Change in Adult ADHD Self Report Scale (ASRS) Symptom Checklist Executive Dysfunction (EFD) Subscale Score
Description: The ASRS is a 31-item questionnaire that assesses the frequency of ADHD symptoms over the past 7 days. Items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The ASRS includes several subscales: an Inattentive (IA) subscale (n = 9), a Hyperactive-Impulsive (HI) subscale (n = 9), an Executive Function Deficits (EFD) subscale (n = 9), and an Emotional Dyscontrol (ED) subscale (n = 4). It also yields a total combined ADHD symptom score. The EFD score ranges from 0-36. Higher scores indicating greater symptom severity.symptoms.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 12.6 (6.2)

10. Secondary Outcome: Change in Adult ADHD Self Report Scale (ASRS) Symptom Checklist Score Overall Emotional Dyscontrol (ED) Subscale Score
Description: The ASRS is a 31-item questionnaire that assesses the frequency of ADHD symptoms over the past 7 days. Items are rated on a 5-point Likert scale ranging from 0 (never) to 4 (very often). The ASRS includes several subscales: an Inattentive (IA) subscale (n = 9), a Hyperactive-Impulsive (HI) subscale (n = 9), an Executive Function Deficits (EFD) subscale (n = 9), and an Emotional Dyscontrol (ED) subscale (n = 4). It also yields a total combined ADHD symptom score. The ED score ranges from 0-36. Higher scores indicating greater symptom severity.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 5.9 (5)

11. Secondary Outcome: Change in 1-Hour Post-Dose Time-Sensitive ADHD Symptom Scale (TASS) Score
Description: 18-item assessment of ADHD symptoms. Each item is rated on a 4-point Likert scale from 0 (not at all) to 3 (severe). The total score is the sum of responses and ranges from 0 to 54; higher scores indicate greater severity of symptoms.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 15
score on a scale | 12.3 (10)

12. Secondary Outcome: Change in 4-Hour Post-Dose TASS Score
Description: as for outcome 11
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 15
score on a scale | 12.6 (10.5)

13. Secondary Outcome: Change in 12-Hour Post-Dose TASS Score
Description: as for outcome 11
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 15
score on a scale | 9.3 (10.5)

14. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 4-Hour Post Dose Score
Description: AMSES is used to assess the smoothness of effect of ADHD medication at specified timepoints throughout the day (4, 6, 8, 10, and 12 hours after dosing). At each timepoint, participants are asked to rate whether the medication's effect feels the same as when they first took it in the morning, using a 5-point Likert scale ranging from 0 (never) to 4 (very often). Higher scores indicate greater smoothness of medication effect.
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 2.86 (0.95)

15. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 6-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 2.64 (0.74)

16. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 8-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 2.07 (0.62)

17. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 10-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 1.64 (0.84)

18. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 12-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 1.21 (1.05)

19. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 4-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 3 (0.88)

20. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 6-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 2.9 (0.66)

21. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 8-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 2.4 (1.08)

22. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 10-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 1.8 (1.19)

23. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 12-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 1.43 (1.16)

24. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 4-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 12
score on a scale | 3.3 (0.78)

25. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 6-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 12
score on a scale | 3.2 (0.72)

26. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 8-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 12
score on a scale | 2.5 (1)

27. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 10-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 12
score on a scale | 1.6 (0.9)

28. Secondary Outcome: Adult ADHD Medication Smoothness of Effect Scale (AMSES) - 12-Hour Post Dose Score
Description: as for outcome 14
Time Frame: Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 12
score on a scale | 1.58 (1.24)

29. Secondary Outcome: AMSES - Overall Smoothness of Effect Scale Score
Description: AMSES is is an assessment of the smoothness of effect of ADHD medication throughout the day following dosing. The overall smoothness of effect scale is a subscale part of the AMSES that asks participants to respond to "How smooth do you think your medication effect is throughout the day?" on a scale from 0 (never) to 100 (very often). The higher the score, the smoother the medication effect is throughout the day.
Time Frame: Week 3
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 69.64 (14.47)

30. Secondary Outcome: AMSES - Overall Smoothness of Effect Scale Score
Description: AMSES is an assessment of the smoothness of effect of ADHD medication throughout the day following dosing. The overall smoothness of effect scale is a subscale part of the AMSES that asks participants to respond to "How smooth do you think your medication effect is throughout the day?" on a scale from 0 (never) to 100 (very often). The higher the score, the smoother the medication effect is throughout the day.
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 14
score on a scale | 75 (21.92)

31. Secondary Outcome: AMSES - Overall Smoothness of Effect Scale Score
Description: as for outcome 30
Time Frame: Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 12
score on a scale | 85.4 (19.82)

32. Secondary Outcome: Change in Behavioral Regulation Index (BRI) T-Score
Description: The Behavioral Regulation Index (BRI) t-score on the BRIEF-A (Behavior Rating Inventory of Executive Function-Adult Version) is a summary measure of an individual's ability to regulate their behavior and emotions, 50 indicates the population mean with a standard deviation of 10. A t-score of 65 or higher indicates difficulties in behavioral regulation.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 15
T-score | 11.9 (12)

33. Secondary Outcome: Change in Metacognition Index (MI) T-Score
Description: The Metacognition Index (MI) t-score on the BRIEF-A (Behavior Rating Inventory of Executive Function-Adult Version) is a measure of executive function that assesses an individual's ability to initiate, plan, organize, self-monitor, and manage their own cognitive processes, 50 indicates the population mean with a standard deviation of 10. A t-score of 65 or higher indicates difficulties with executive function related to planning, organization, and cognitive self-regulation.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 15
T-score | 22.1 (15.3)

34. Secondary Outcome: Change in Global Executive Composite (GEC) T-score
Description: The Global Executive Composite (GEC) t-score on the BRIEF-A (Behavior Rating Inventory of Executive Function-Adult Version) is a summary measure of overall executive function, 50 indicates the population mean with a standard deviation of 10. A t-score of 65 or higher indicates difficulties with executive function in daily life.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 15
T-score | 19.2 (14.3)

35. Secondary Outcome: Change in Clinical Global Impression-Severity (CGI-S) Scale Score
Description: 1-item clinician-rated assessment of the severity of a subject's mental illness. The severity of illness is rated as follows: 0 (not assessed), 1 (normal, not at all ill), 2 (borderline mentally ill), 3 (mildly ill), 4 (moderately ill), 5 (markedly ill), 6 (severely ill), 7 (among the most extremely ill subjects). The total score is the numerical ranking provided by the clinician.
Time Frame: Week 2, Week 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adult ADHD Patients
Number analyzed (Participants) | 15
score on a scale | 1.7 (1)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Adult ADHD Patients
All-Cause Mortality (participants affected / at risk) | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 13/29
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adult ADHD Patients (N=29)
Pain in fingers and hands (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 9
Nausea (Gastrointestinal disorders) | 6
Insomnia (Nervous system disorders) | 5
Upset stomach /loose stool (Gastrointestinal disorders) | 2
Metallic taste (Nervous system disorders) | 1
muscle stiffness (Musculoskeletal and connective tissue disorders) | 1
Gastroenteritis (Gastrointestinal disorders) | 1
anxiety (Psychiatric disorders) | 7
intermittent irritability (Nervous system disorders) | 1
Menstrual cramps (Reproductive system and breast disorders) | 1
common cold (Infections and infestations) | 2
fatigue (Nervous system disorders) | 4
dry mouth (Gastrointestinal disorders) | 2
decreased appetite (Gastrointestinal disorders) | 2
wisdom teeth pain (General disorders) | 1
Increased heart rate (Cardiac disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/01/NCT06000501/Prot_SAP_000.pdf